CLINICAL TRIAL: NCT00545025
Title: Safety and Immunogenicity of a Second Vaccination With GSK Biologicals' Influenza Vaccine GSK1247446A in Subjects 18-60 Years Previously Vaccinated in Study 108656
Brief Title: Revaccination With Influenza Vaccine GSK1247446A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110674; 2007-002783-10 (EudraCT Number)
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Influenza; Influenza, Human
Keywords: Influenza; Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (2):
- GSK1247446A Group (Experimental): Subjects aged between 18 and 60 years, having previously received one dose of the AS03-adjuvanted GSK1247446A vaccine in the primary study NCT00374842, received a single dose of GSK1247446A vaccine adjuvanted with a half dose of AS03 adjuvant at Day 0 of the current follow-up study NCT00545025. The vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm. Subjects in this group originated from either the GSK1247446A Formulation 1 or GSK1247446A Formulation 2 groups in study NCT00374862.
  Interventions: Biological: Influenza Vaccine GSK1247446A
- Fluarix Group (Active Comparator): Subjects aged between 18 and 60 years, having previously received one dose of Fluarix™ vaccine during the primary study NCT00374842, received one dose of Fluarix™ vaccine at Day 0 of the current follow-up study NCT00545025. The vaccine was administered intramuscularly, in the deltiod region of the non-dominant arm. Subjects in this group originated from the Fluarix Group in study NCT00374862.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Influenza Vaccine GSK1247446A — Single dose, Intramuscular injection
  Arms: GSK1247446A Group
Biological: Fluarix™ — Single dose, Intramuscular injection
  Arms: Fluarix Group

SUMMARY:
The protocol is designed to demonstrate the safety of influenza vaccine GSK1247446A after revaccination.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18-60 years old at the time of vaccination, who previously participated in 108656 clinical trial.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period
* Previous vaccination against influenza since January 2007.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Administration of immunoglobulins and/or any blood products within three months preceding the dose of study vaccine or planned administration during the study period.
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of confirmed influenza infection within the last 12 months.
* Pregnancy.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute disease at the time of enrolment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 243 (Actual)
Dates: Start 2007-10-15 (Actual); Primary Completion 2007-12-12 (Actual); Study Completion 2007-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 110674 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110674 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110674 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110674 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110674 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110674 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled and vaccinated in this NCT00545025 follow-up previously participated in the NCT00374842 study, wherein they were vaccinated with either the GSK1247446A or Fluarix™ vaccines.
Pre-assignment Details: Subjects were allocated to study groups based on their vaccination course in the NCT00374842 primary study, so as to receive a re-vaccination dose of the vaccine previously administered.
Groups:
- Fluarix Group: Subjects aged between 18 and 60 years, having previously received one dose of Fluarix™ vaccine during the primary study NCT00374842, received one dose of Fluarix™ vaccine at Day 0 of the current follow-up study NCT00545025. The vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm. Subjects in this group originated from the Fluarix Group in study NCT00374862.
Period: Overall Study
Arm/Group | GSK1247446A Group | Fluarix Group
Started | 160 | 83
Completed | 160 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1247446A Group | Fluarix Group | Total
Number analyzed (Participants) | 160 | 83 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (13.66) | 40.9 (13.66) | 39.9 (13.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 44 | 142
  Male | 62 | 39 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, pain, redness and swelling at injection site. Any = incidence of a particular symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal everyday activity. Grade 3 redness/swelling/ecchymosis = redness/swelling/ecchymosis spreading beyond 50 millimeters (mm) of the injection site. All solicited local symptoms assessed were considered by the investigator as related to study vaccination.
Time Frame: During a 7-day (Days 0-6) follow-up period after re-vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 160 | 83
Subjects
  Any Ecchymosis | 8 | 5
  Ecchymosis > 50mm | 1 | 2
  Any Pain | 143 | 57
  Grade 3 Pain | 9 | 2
  Any Redness | 24 | 10
  Redness > 50mm | 2 | 1
  Any Swelling | 29 | 13
  Swelling > 50mm | 4 | 2

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [oral temperature equal to or above ≥ 37.5 degrees Celsius (°C)], headache, myalgia, nausea and shivering. Any = incidence of a particular symptom regardless of grade intensity or relationship with the study vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0°C. Related = symptom considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During a 7-day (Days 0-6) follow-up after re-vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 160 | 83
Subjects
  Any Arthralgia | 28 | 5
  Grade 3 Arthralgia | 3 | 0
  Related Arthralgia | 26 | 5
  Any Fatigue | 72 | 12
  Grade 3 Fatigue | 7 | 2
  Related Fatigue | 71 | 10
  Fever ≥37.5°C | 27 | 2
  Fever >39.0°C | 0 | 0
  Related Fever | 27 | 2
  Any Headache | 65 | 18
  Grade 3 Headache | 6 | 1
  Related Headache | 61 | 16
  Any Myalgia | 56 | 8
  Grade 3 Myalgia | 4 | 0
  Related Myalgia | 52 | 8
  Any Nausea | 23 | 4
  Grade 3 Nausea | 0 | 0
  Related Nausea | 21 | 3
  Any Shivering | 39 | 3
  Grade 3 Shivering | 4 | 0
  Related Shivering | 39 | 2

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = unsolicited AE that prevented normal activity. Related = unsolicited AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 30-day (Days 0-29) follow-up period after re-vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 160 | 83
Subjects
  Any AEs | 69 | 31
  Grade 3 AEs | 16 | 10
  Related AEs | 35 | 8

4. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Related = SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Days 0-30)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 160 | 83
Subjects
  Any SAEs | 0 | 1
  Related SAEs | 0 | 0

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 3 influenza strains assessed were A/Solomon Islands (A/SOL), A/Wisconsin (A/WIS) and B/Malaysia (B/MAL). The seropositivity cut-off assay was 1:10.
Time Frame: At Days 0 and 21
Population: The analysis was based on the according-to-protocol (ATP) Cohort for immunogenicity, which included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after revaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 159 | 82
Titer
  A/SOL, Day 0 [N=158, 82] | 41.0 [32.2 to 52.3] | 43.0 [29.7 to 62.1]
  A/SOL, Day 21 [N=159, 82] | 162.4 [140.0 to 188.4] | 127.2 [97.2 to 166.5]
  A/WIS, Day 0 [N=158, 82] | 83.2 [71.3 to 97.1] | 78.9 [61.2 to 101.8]
  A/WIS, Day 21 [N=159, 82] | 191.7 [171.7 to 214.0] | 147.0 [121.6 to 177.6]
  B/MAL, Day 0 [N=158, 82] | 107.3 [89.3 to 128.8] | 75.7 [57.6 to 99.4]
  B/MAL, Day 21 [N=159, 82] | 334.2 [296.0 to 377.4] | 199.3 [164.5 to 241.5]

6. Secondary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 3 influenza strains assessed were A/Solomon Islands (A/SOL), A/Wisconsin (A/WIS) and B/Malaysia (B/MAL).
Time Frame: At Day 21
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 159 | 82
Subjects
  A/SOL | 73 | 30
  A/WIS | 40 | 13
  B/MAL | 61 | 23

7. Secondary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 3 influenza strains assessed were A/Solomon Islands (A/SOL), A/Wisconsin (A/WIS) and B/Malaysia (B/MAL).
Time Frame: At Day 0 and 21
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 159 | 82
Subjects
  A/SOL, Day 0 [N=158, 82] | 87 | 45
  A/SOL, Day 21 [159, 82] | 155 | 75
  A/WIS, Day 0 [N=158, 82] | 139 | 69
  A/WIS, Day 21 [N=159, 82] | 159 | 80
  B/MAL, Day 0 [N=158, 82] | 133 | 67
  B/MAL, Day 21 [N=159, 82] | 159 | 82

8. Secondary Outcome: Seroconversion Factor for HI Antibodies Against 3 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 3 influenza strains assessed were A/Solomon Islands (A/SOL), A/Wisconsin (A/WIS) and B/Malaysia (B/MAL).
Time Frame: At Day 21
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK1247446A Group | Fluarix Group
Number analyzed (Participants) | 158 | 82
Fold increase
  A/SOL | 3.9 [3.3 to 4.8] | 3.0 [2.3 to 3.8]
  A/WIS | 2.3 [2.1 to 2.6] | 1.9 [1.6 to 2.2]
  B/MAL | 3.1 [2.7 to 3.6] | 2.6 [2.2 to 3.2]

ADVERSE EVENTS:
Time Frame: Reports for solicited local and general symptoms were collected during the 7 (Days 0-6) days post revaccination. Reports for AEs were collected during the 30 (Days 0-29) days post revaccination and SAEs during the whole study period (Day 0 - Month 1).
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Groups:
- GSK1247446A Group: Subjects aged between 18 and 60 years, having previously received one dose of the AS03-adjuvanted GSK1247446A vaccine adjuvanted with a full dose of AS03-adjuvant in the primary study NCT00374842, received a single dose of GSK1247446A vaccine adjuvanted with a half dose of AS03- adjuvant at Day 0 of the current follow-up study NCT00545025. The vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm. Subjects in this group originated from either the GSK1247446A Formulation 1 or GSK1247446A Formulation 2 groups in study NCT00374862.
Arm/Group | GSK1247446A Group | Fluarix Group
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/160 | 1/83
Other Adverse Events (participants affected / at risk) | 143/160 | 57/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A Group (N=160) | Fluarix Group (N=83)
Cerebrovascular accident (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A Group (N=160) | Fluarix Group (N=83)
Nasopharyngitis (Infections and infestations) | 15 | 12
Headache (Nervous system disorders) | 8 | 3 — Headache was reported as an unsolicited adverse event (AE).
Diarrhoea (Gastrointestinal disorders) | 9 | 1
Arthralgia (General disorders) | 28 | 5
Fatigue (General disorders) | 72 | 12
Fever (General disorders) | 27 | 2 — Fever was defined as oral temperature ≥ 37.5 degrees Celsius (°C)
Headache (General disorders) | 65 | 18
Myalgia (General disorders) | 56 | 8
Nausea (General disorders) | 23 | 4
Shivering (General disorders) | 39 | 3
Ecchymosis (General disorders) | 8 | 5
Pain (General disorders) | 143 | 57
Redness (General disorders) | 24 | 10
Swelling (General disorders) | 29 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.